CLINICAL TRIAL: NCT07308873
Title: Individual Differences in Gait and Osteoarthritis Pain
Acronym: INDIGO
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Benedict Alter, Assistant Professor, University of Pittsburgh
Other Study IDs: STUDY25080027; 1R01AR086796-01 (NIH)
Record Dates: First submitted 2025-12-26; First posted 2025-12-30 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis (OA); Chronic Pain; Chronic Knee Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic knee pain with knee osteoarthritis: Adults 45-80 years old who have moderately severe knee osteoarthritis. They must have experienced knee pain for greater than 6 months and rate their daily knee pain at >3 on a 0-10 numeric rating scale.

SUMMARY:
The goal of this observational study is to look at inter-individual differences in knee osteoarthritis (OA) walking pain and performance. The main questions this study aims to answer are:

Why do some people with knee osteoarthritis have more severe disabling pain than others, even though the degenerative changes in their knees are similar?

What are the factors that contribute to walking pain in people with knee osteoarthritis?

Participants will complete surveys, perform physical function tasks, get a knee X-ray and MRI, undergo non-invasive brain imaging, and undergo sensory testing.

DETAILED DESCRIPTION:
This observational study will identify biopsychosocial factors that contribute to inter-individual differences in walking pain and pain limiting walking with the hypothesis that neural processes play a key role. This study's objective is to elucidate "whole person" biopsychosocial mechanisms of movement-evoked pain and pain limitations on function in knee OA, helping to determine why some patients have severe disabling pain while others do not despite similar degenerative changes of the knee joint. Three hundred participants with knee OA will undergo a comprehensive data collection over two study visits, including surveys, exercise tasks, non-invasive brain and joint imaging, and biomechanics assessments during mobility. Using advanced analysis, this dataset will be used to identify factors contributing to walking-evoked pain and functional limitations in knee osteoarthritis.These results will identify new therapeutic targets to maintain or improve physical activity in patients with knee osteoarthritis, leading to better outcomes of physical therapy and improved overall health and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Knee pain for greater than 6 months.
* Moderate-to-severe knee pain (>3/10) due to osteoarthritis, as defined by American College of Rheumatology and EULAR diagnostic criteria, on >50% of days in the past month.
* KL grade 2-4 indicating significant degenerative changes on knee X-ray.
* 45-80 years old

Exclusion Criteria:

* Inflammatory arthritis (e.g. rheumatoid arthritis).
* More intense pain due to another chronic pain syndrome (e.g. fibromyalgia, hip osteoarthritis)
* Significant pain or weakness in the lower extremities due to a neurological condition (e.g. lumbar radiculopathy, paresis due to stroke)
* Acute pain that is more intense than knee osteoarthritis pain
* Current routine use of more than 15 mg oral morphine equivalents per day (use of <15 mg OME does not exclude the participant).
* Recent new medication, exercise, behavioral, or complementary and integrative treatment started in the last month. Stable use of these treatments for greater than 1 month does not exclude the participant.
* Recent intra-articular injection of steroid or other agent (greater than 1 month does not exclude the participant)
* Recent knee radiofrequency ablation (greater than 3 months does not exclude the participant)
* Recent knee arthroscopic surgery (greater than 3 months does not exclude the participant)
* History of knee replacement or open knee surgery on the index knee, defined as the more painful knee on average over the last month.
* Inability to walk or climb stairs without significant assistance (e.g. a one-person assist, use a wheel chair; however, the use of a cane does not exclude the participant).
* Inability to participate in study procedures (e.g. cognitive impairment limiting ability to understand directions, inability to understand and read English)
* Uncontrolled or unstable medical disorder preventing participation in study procedures
* History of brain surgery
* Tattoos on sensory testing sites
* Pregnancy
* Breastfeeding
* Inability to under knee MRI scan due to incompatible devices or foreign bodies.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample includes participants with knee osteoarthritis of at least moderate pain severity and radiographic evidence of significant knee joint degeneration. Participants will be recruited from research registries (Pitt CTSI Pitt+Me) and clinics with a high volume of knee osteoarthritis patients, including orthopedic and pain management clinics. Eligibility criteria are designed to study knee osteoarthritis pain around the time of walking. Therefore, some comorbidities and pain conditions are allowed if knee osteoarthritis is the primary pain condition, but other painful conditions are not allowed due to a significant confounding effect on the study. Concurrent knee interventions, such as injections, have different expected time courses of treatment effects. The exclusion criteria timepoints for each intervention are meant to enroll participants at a relatively stable periods of time after the interventions, so that pain and function do not change dramatically across Study Visits.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-07 (Actual); Primary Completion 2030-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
6 minute walk test pain intensity | 6 minutes
  Pain intensity on numeric rating scale (0-10) during and around the time of the 6-minute walk test.

SECONDARY OUTCOMES:
Distance walked in the 6-minute walking test | 6 minutes
  Distance walked during 6 minute walking task

OTHER OUTCOMES:
Quantitative sensory testing | 2-3 hours
  Responses to quantitative sensory tests that assess sensation of painful and non-painful stimuli. The stimuli are calibrated and carefully controlled with safety measures to prevent tissue damage.
Physical function performance and pain | 2-3 hours
  A battery of standardized physical function tests including a stair climb test, fast-paced walk test, balance test, and sit-to-stand test, will be done to measure physical performance. Outcome measurements include the time to complete the test, distance walked, and number of repetitions. Pain intensity is reported on the numeric rating scale (0-10) during this battery of tests.
Brain imaging | 2-3 hours
  Brain activity will be measured non-invasively using functional near-infrared spectroscopy
Biomechanics during physical activity | 3-4 hours
  Aspects of body movement will be measured non-invasively during physical performance tests, including the 6-minute walk test
Multidimensional pain assessment | 1 hour
  Multidimensional aspects of chronic pain will be measured through written surveys and a semi-structured clinical evaluation.
Knee MRI | 1 hour
  Structural changes of the knee will be measured, including the use of standard scoring systems.

CONTACTS AND LOCATIONS:
Overall Officials: Benedict Alter, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Pain Medicine at Centre Commons, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared in accordance with NIH HEAL regulatory requirements.
Supporting Information: Study Protocol, ICF
Time Frame: IPD will be shared in accordance with NIH HEAL requirements, meaning that IPD will be made publicly available after the publication of results.
Access Criteria: IPD will be publicly available.